CLINICAL TRIAL: NCT00944021
Title: A Phase II Dose Ranging Trial to Evaluate the Extended Early Bactericidal Activity, Safety, Tolerability, and Pharmacokinetics of PA-824 in Adult Participants With Newly Diagnosed, Uncomplicated, Smear-Positive, Pulmonary Tuberculosis
Brief Title: Evaluation of Early Bactericidal Activity in Pulmonary Tuberculosis (CL-010)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Global Alliance for TB Drug Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PA-824-CL-010
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Results first posted 2016-03-09 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Pulmonary Tuberculosis
Keywords: Early Bactericidal Activity; EBA; Pulmonary Tuberculosis; PA-824; pretomanid
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — pretomanid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- PA-824 50 mg/qd (Experimental)
  Interventions: Drug: PA-824
- PA-824 100mg/qd (Experimental)
  Interventions: Drug: PA-824
- PA-824 150mg/qd (Experimental)
  Interventions: Drug: PA-824
- PA-824 200mg/qd (Experimental)
  Interventions: Drug: PA-824
- Rifafour e-275mg (Active Comparator)
  Interventions: Drug: Rifafour e-275 mg

INTERVENTIONS:
Drug: PA-824 — 50mg
  Arms: PA-824 50 mg/qd
Drug: PA-824 — 100mg
  Arms: PA-824 100mg/qd
Drug: PA-824 — 150 mg
  Arms: PA-824 150mg/qd
Drug: Rifafour e-275 mg — 275 mg
  Arms: Rifafour e-275mg
Drug: PA-824 — 200 mg
  Arms: PA-824 200mg/qd

SUMMARY:
The trial will evaluate the extended bactericidal activity of 14 consecutive days of oral administration of PA-824 at 50, 100, 150 and 200 mg per day in adult patients with newly diagnosed, uncomplicated, smear positive tuberculosis (TB). A control group will receive standard TB treatment.

DETAILED DESCRIPTION:
The planned sample size of 15 participants per treatment group is in keeping with other Phase II trials of this type and accounts for the possibility of up to 3 drop-outs per arm, which based on previous studies of this type conducted at these sites, represents a conservative estimate of the expected drop-out rate.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* Body weight between 40 and 90 kg, inclusive.
* Newly diagnosed, previously untreated, uncomplicated, sputum smear-positive, pulmonary TB.
* A chest X-ray compatible with TB.
* Sputum positive
* Adequate volume of sputum
* Female participants of childbearing potential negative serum pregnancy and agree to use birth control
* Male participants must agree to use contraception throughout participation in the trial and for 12 weeks after last dose.

Exclusion Criteria:

* Poor general condition
* Rifampicin-resistant and/or Isoniazid-resistant
* MTB Treatment received within the 3 months prior
* Allergy to the IMP or related substances
* Evidence of extrathoracic TB
* A history of previous TB
* Evidence of serious lung conditions other than TB or uncontrolled obstructive bronchial disease
* History of lens opacity or evidence of lens opacity on slit lamp ophthalmologic examination
* Any evidence of renal impairment
* For males, any evidence or history of abnormality in the reproductive system
* History and/or presence (or evidence) of neuropathy or epilepsy.
* Clinically relevant changes in the ECG
* A history of or current clinically relevant cardiovascular disorder
* Concomitant use of any drug known to prolong QTc interval
* Diabetics using insulin
* Evidence of clinically significant metabolic, gastrointestinal, neurological, psychiatric or endocrine diseases, malignancy, or other abnormalities (other than the indication being studied).
* Any diseases or conditions in which the use of the standard TB drugs or any of their components is contra-indicated, including but not limited to allergy to any TB drug, their component or to the IMP.
* Any disease or conditions in which any of the medicinal products listed in the section pertaining to prohibited medication is used.
* alcohol or drug abuse
* Administration of an IMP prior to Visit 1, within 5 half-lives for that IMP if known. If the half-life of the IMP is unknown within 1 month.
* Pregnant, breast-feeding, or planning to conceive or father a child within twelve weeks of cessation of treatment for males and within one week of cessation of treatment for females.
* Use of any drugs or substances within 30 days prior to dosing known to be strong inhibitors or inducers of cytochrome P450 enzymes
* Any therapeutic agents known to alter any major organ function (e.g., barbiturates, opiates, phenothiazines, cimetidine) within 30 days prior to dosing.
* glucocorticoids within one year prior to dosing.
* HIV infection with helper/inducer T lymphocyte (CD4 cell) count of less than or equal to 300x10-6/L.
* Receiving antiretroviral therapy (ART).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2009-08; Primary Completion 2010-01 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Diacon, MD, Principal Investigator — Karl Bremer Hospital; Rodney Dawson, MD, Principal Investigator — University of Cape Town Lung Institute

REFERENCES:
- [Result] Diacon AH, Dawson R, du Bois J, Narunsky K, Venter A, Donald PR, van Niekerk C, Erondu N, Ginsberg AM, Becker P, Spigelman MK. Phase II dose-ranging trial of the early bactericidal activity of PA-824. Antimicrob Agents Chemother. 2012 Jun;56(6):3027-31. doi: 10.1128/AAC.06125-11. Epub 2012 Mar 19. PMID 22430968

RESULTS

PARTICIPANT FLOW:
Groups:
- PA-824 50 mg/qd: PA-824 : 50mg oral tablet
- PA-824 100mg/qd: PA-824 : 100mg oral tablet
- PA-824 150mg/qd: PA-824 : 150 mg oral tablet
- PA-824 200mg/qd: PA-824 : 200 mg oral tablet
- Rifafour e-275mg: Rifafour e-275 mg : A once daily dose dependent on the patients weight 30 to 37 kg - 2 tablets, 38 to 54 kg - 3 tablets, 55 to 70 kg - 4 tablets or 71 kg and over - 5 tablets).
Period: Overall Study
Arm/Group | PA-824 50 mg/qd | PA-824 100mg/qd | PA-824 150mg/qd | PA-824 200mg/qd | Rifafour e-275mg
Started | 15 | 15 | 15 | 16 | 8
Completed | 14 | 15 | 15 | 16 | 8
Not Completed | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PA-824 50 mg/qd | PA-824 100mg/qd | PA-824 150mg/qd | PA-824 200mg/qd | Rifafour e-275mg | Total
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 8 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 15 | 16 | 8 | 69
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (9.76) | 29.6 (9.28) | 26.9 (8.91) | 25.3 (6.18) | 33.3 (14.09) | 28.6 (9.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 8 | 9 | 2 | 34
  Male | 7 | 8 | 7 | 7 | 6 | 35
Region of Enrollment [Number; unit: participants]
  South Africa | 15 | 15 | 15 | 16 | 8 | 69

OUTCOME MEASURES:

1. Primary Outcome: Early Bactericidal Activity (EBA) Measured as the Mean Rate of Reduction of log10 Colony Forming Units (CFU) of M. Tuberculosis Per ml Sputum on Solid Medium Over Time (Days 0-14).
Time Frame: 14 consecutive days of treatment
Population: All randomized subjects. Some of the EBA values could not be calculated due to missing results. The analysis population is the number of patients for whom the results were available for this time period and therefore for whom the relevant EBA could be calculated.
Measure: Mean (Standard Deviation); unit: log10CFU/ml/day
Arm/Group | PA-824 50 mg/qd | PA-824 100mg/qd | PA-824 150mg/qd | PA-824 200mg/qd | Rifafour e-275mg
Number analyzed (Participants) | 12 | 15 | 14 | 14 | 8
log10CFU/ml/day | 0.063 (0.058) | 0.091 (0.073) | 0.078 (0.074) | 0.112 (0.070) | 0.177 (0.042)

2. Secondary Outcome: Early Bactericidal Activity (EBA) Measured as the Mean Rate of Reduction of log10 Colony Forming Units (CFU) of M. Tuberculosis Per ml Sputum on Solid Medium Over Time (Days 0-2).
Time Frame: Two consecutive days of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log10CFU/ml/day
Arm/Group | PA-824 50 mg/qd | PA-824 100mg/qd | PA-824 150mg/qd | PA-824 200mg/qd | Rifafour e-275mg
Number analyzed (Participants) | 14 | 15 | 15 | 14 | 8
log10CFU/ml/day | 0.093 (0.211) | 0.111 (0.332) | -0.009 (0.290) | 0.160 (0.255) | 0.470 (0.316)

3. Secondary Outcome: Early Bactericidal Activity (EBA) Measured as the Mean Rate of Reduction of log10 Colony Forming Units (CFU) of M. Tuberculosis Per ml Sputum on Solid Medium Over Time (Days 2-14).
Time Frame: Days 2-14 of 14 consecutive days of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log10CFU/ml/day
Arm/Group | PA-824 50 mg/qd | PA-824 100mg/qd | PA-824 150mg/qd | PA-824 200mg/qd | Rifafour e-275mg
Number analyzed (Participants) | 12 | 15 | 14 | 14 | 8
log10CFU/ml/day | 0.059 (0.060) | 0.088 (0.085) | 0.096 (0.98) | 0.104 (0.083) | 0.128 (0.070)

4. Secondary Outcome: Rate of Change in Increased Time to Sputum Culture Positivity (TTP)(Hours) in Liquid Culture Media (Days 0-14).
Time Frame: Fourteen consecutive days of treatment
Population: All randomized subjects. Some of the TTP values could not be calculated due to missing results. The population is the number of patients for whom the results were available for this time period and therefore for whom the relevant TTP could be calculated.
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | PA-824 50 mg/qd | PA-824 100mg/qd | PA-824 150mg/qd | PA-824 200mg/qd | Rifafour e-275mg
Number analyzed (Participants) | 13 | 14 | 15 | 16 | 8
hours/day | 2.621 (2.534) | 4.969 (3.644) | 4.633 (3.687) | 4.640 (3.447) | 13.364 (3.979)

5. Secondary Outcome: Rate of Change in Increased Time to Sputum Culture Positivity (TTP)(Hours) in Liquid Culture Media (Days 0-2).
Time Frame: Two consecutive days of treatment
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | PA-824 50 mg/qd | PA-824 100mg/qd | PA-824 150mg/qd | PA-824 200mg/qd | Rifafour e-275mg
Number analyzed (Participants) | 15 | 14 | 15 | 13 | 8
hours/day | 1.483 (8.153) | -1.345 (8.586) | 4.867 (12.755) | 3.096 (8.202) | 37.016 (5.639)

6. Secondary Outcome: Rate of Change in Increased Time to Sputum Culture Positivity (TTP)(Hours) in Liquid Culture Media (Days 2-14).
Time Frame: Days 2-14 of 14 consecutive days of treatment
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | PA-824 50 mg/qd | PA-824 100mg/qd | PA-824 150mg/qd | PA-824 200mg/qd | Rifafour e-275mg
Number analyzed (Participants) | 13 | 15 | 15 | 13 | 8
hours/day | 2.958 (2.652) | 5.744 (3.973) | 4.594 (5.035) | 5.391 (3.608) | 9.422 (4.367)

7. Secondary Outcome: Pharmacokinetics- Maximum Observed Plasma Concentration (Cmax) (Day 1).
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 12, 16, and 24 hours post-dose on Day 1 of treatment
Population: All PA-824 patients who received at least one administration of the investigational drug, had at least one measured concentration after the start of treatment for at least one PK analysis and had no major events affecting the integrity of the PK data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PA-824 50 mg/qd | PA-824 100mg/qd | PA-824 150mg/qd | PA-824 200mg/qd
Number analyzed (Participants) | 15 | 15 | 15 | 16
ng/mL | 465.3 (150.6) | 662.3 (167.8) | 994.7 (305.7) | 1183.0 (382.5)

8. Secondary Outcome: Pharmacokinetics- Area Under the Plasma Concentration Time Curve From Zero to Infinity (AUC 0 to Infinity) (Day 1).
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 12, 16, and 24 hours post-dose on Day 1 of treatment
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng * hour/mL
Arm/Group | PA-824 50 mg/qd | PA-824 100mg/qd | PA-824 150mg/qd | PA-824 200mg/qd
Number analyzed (Participants) | 15 | 15 | 15 | 16
ng * hour/mL | 11923.94 (4512.94) | 18408.59 (7665.35) | 28654.83 (10924.23) | 38485.04 (16606.96)

9. Secondary Outcome: Pharmacokinetics- Terminal Elimination Phase Half-life (t1/2) (Day 1).
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 12, 16, and 24 hours post-dose on Day 1 of treatment
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PA-824 50 mg/qd | PA-824 100mg/qd | PA-824 150mg/qd | PA-824 200mg/qd
Number analyzed (Participants) | 15 | 15 | 15 | 16
hours | 16.142 (5.501) | 18.597 (9.459) | 19.005 (7.349) | 21.092 (6.490)

10. Secondary Outcome: Pharmacokinetics-Maximum Observed Plasma Concentration (Cmax) (Day 14).
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 12,16, 24, and 30 hours post-dose on Day 14 of 14 consecutive days of treatment
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PA-824 50 mg/qd | PA-824 100mg/qd | PA-824 150mg/qd | PA-824 200mg/qd
Number analyzed (Participants) | 15 | 15 | 15 | 16
ng/mL | 777.3 (250.7) | 1116.5 (357.4) | 1543.9 (511.4) | 2223.8 (734.5)

11. Secondary Outcome: Pharmacokinetics- Terminal Elimination Phase Half-life (t1/2) (Day 14).
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 12, 16, 24 and 30 hours post-dose on Day 14 of 14 consecutive days of treatment
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | PA-824 50 mg/qd | PA-824 100mg/qd | PA-824 150mg/qd | PA-824 200mg/qd
Number analyzed (Participants) | 15 | 15 | 15 | 16
hour | 18.645 (5.394) | 19.274 (10.249) | 20.207 (5.288) | 23.811 (8.067)

ADVERSE EVENTS:
Time Frame: 180 days
Description: Adverse events were collected from the time a patient signed the informed consent until day 29. From day 29 through day 180, only opthalmologic related adverse events and serious adverse events were collected. Data reported are treatment-emergent adverse events.
Arm/Group | PA-824 50 mg/qd | PA-824 100mg/qd | PA-824 150mg/qd | PA-824 200mg/qd | Rifafour e-275mg
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/15 | 0/15 | 1/16 | 0/8
Other Adverse Events (participants affected / at risk) | 10/15 | 5/15 | 5/15 | 7/16 | 4/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PA-824 50 mg/qd (N=15) | PA-824 100mg/qd (N=15) | PA-824 150mg/qd (N=15) | PA-824 200mg/qd (N=16) | Rifafour e-275mg (N=8)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 | 0 (0) | 0 (0) | 1 | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PA-824 50 mg/qd (N=15) | PA-824 100mg/qd (N=15) | PA-824 150mg/qd (N=15) | PA-824 200mg/qd (N=16) | Rifafour e-275mg (N=8)
Bundle branch block left (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 1 | 0 | 0 | 0
Lenticular opacities (Eye disorders) | 0 | 0 | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1
Chills (General disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Heart rate increased (Investigations) | 0 | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Euphoric mood (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 3 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other